CLINICAL TRIAL: NCT04588064
Title: Comparison of 18F-FDG and 68Ga-FAPI PET/CT in Patients with Lung Adenocarcinoma
Brief Title: 18F-FDG and 68Ga-FAPI PET/CT in Lung Adenocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KYZ2017-001
Record Dates: First submitted 2020-09-13; First posted 2020-10-19 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Lung Adenocarcinoma; 18F-FDG; 68Ga-FAPI; PET/CT
Keywords: Lung Adenocarcinoma; FDG; FAPI; PET/CT
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Intervention Model Description: Participants with lung adenocarcinoma undergo contemporaneous 68Ga-FAPI and 18F-FDG PET/CT for tumor staging before treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18F-FDG PET/CT scan (Experimental): Each subject receives a single intravenous injection of 18F-FDG, and undergo PET/CT imaging within the specified time.
  Interventions: Diagnostic Test: 68Ga-FAPI PET/CT scan

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI PET/CT scan — Each subject receives a single intravenous injection of 68Ga-FAPI, and undergo PET/CT imaging within the specified time.

SUMMARY:
To evaluate the potential usefulness of 68Ga-FAPI positron emission tomography/computed tomography (PET/CT) for the diagnosis of primary and metastatic lesions in lung adenocarcinoma, compared with 18F-FDG PET/CT.

DETAILED DESCRIPTION:
Participants with lung adenocarcinoma underwent contemporaneous 18F-FDG and 68Ga-FAPI PET/CT for an initial assessment. Tumor uptake was quantified by the maximum standard uptake value (SUVmax). The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 18F-FDG and 68Ga-FAPI PET/CT were calculated and compared to evaluate the diagnostic efficacy. In addition, the investigators further investigate the performance of 68Ga-FAPI PET/CT for differentiating invasive adenocarcinoma from adenocarcinoma in situ (pre-invasive lesion) or minimally invasive adenocarcinoma in participants with solitary ground-glass opacity nodules.

ELIGIBILITY:
Inclusion Criteria:

* (i) aged ≥ 18 years, with newly detected GGNs ≤ 3 cm on LDCT and suspected to be lung cancer, and with no prior treatment;
* (ii) who accepted undergoing paired 18F-FDG and 68Ga-FAPI-46 PET/CT, with completion within one week of each other;
* (iii) with planned surgical resection within one month after PET/CT examinations;
* (iv) with an ability to provide informed consent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

* (i) without surgical treatment;
* (ii) receiving antitumor treatment prior to surgery;
* (iii) whose postoperative pathology revealed adenocarcinoma beyond stage IA or benign pulmonary lesions;
* (iv) with concurrent diagnosis of other malignant tumors;
* (v) with poor image quality or lesions difficult to measure.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Cut-off value of SUVmax | 30 days
  Using the cut-off value of SUVmax derived from 68Ga-FAPI-46 PET to distinguish IAC from pre-invasive lesions (including atypical adenomatous hyperplasia (AAH), adenocarcinoma in situ (AIS), and minimally invasive adenocarcinoma (MIA)) in GGNs.

SECONDARY OUTCOMES:
The area under the receiver operating characteristic (ROC) curve (AUC), accuracy, sensitivity, specificity, p-value [indicating accuracy exceeding the No-Information Rate], and kappa value | 30 days
  Based on clinical features (age, sex, smoking history) and PET/CT parameters (including SUVmax, TBR, CT value), calculate the diagnostic performance. Based on 68Ga-FAPI-46 PET/CT radiomics features, calculate the diagnostic performance and explain the most significant predictors.

CONTACTS AND LOCATIONS:
Overall Officials: Long Sun, PhD, Study Director — The First Affiliated Hospital of Xiamen University, Fujian, China
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruan D, Shi S, Guo W, Pang Y, Yu L, Cai J, Wu Z, Wu H, Sun L, Zhao L, Chen H. Evaluation of locoregional invasiveness of early lung adenocarcinoma manifesting as ground-glass nodules via [68Ga]Ga-FAPI-46 PET/CT imaging. Eur J Nucl Med Mol Imaging. 2025 Nov;52(13):4788-4805. doi: 10.1007/s00259-025-07361-5. Epub 2025 May 24. PMID 40411546